CLINICAL TRIAL: NCT02503631
Title: Stool Sample Collection Protocol for Development of Screening Test for Colorectal Cancer and Other Digestive Tract Cancers
Status: Terminated | Type: Observational
Why Stopped: Changes in development plan
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-02
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Colorectal Cancer
Keywords: Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Provide anonymous, clinically characterized specimens and blood samples for bio-repository for future colorectal cancer-related test development.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Subjects will be men and women, 40-90 years of age, inclusive, each with a colonoscopic biopsy-based diagnosis of colorectal cancer (CRC) and/or a pre-malignant colorectal lesion with large enough residual lesion to require subsequent surgical excision or complex colonoscopic polypectomy.
  Interventions: Device: Stool Sample Collection Kit

INTERVENTIONS:
Device: Stool Sample Collection Kit — Stool sample collection kit

SUMMARY:
The primary objective of this study is to obtain de-identified, clinically characterized, stool and plasma specimens for use in assessing new markers for the detection of neoplasms of the digestive tract.

DETAILED DESCRIPTION:
This is a multi-site, prospective sample collection study. Subjects will be men and women, 40-90 years of age, inclusive, each with a colonoscopic biopsy-based diagnosis of CRC and/or a pre-malignant colorectal lesion with large enough residual lesion to require subsequent surgical excision or complex colonoscopic polypectomy.

One stool sample from approximately 300 subjects will be collected in this study. A blood sample will also be collected from subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 40-90 years of age, inclusive.
* Subject has a diagnosis of CRC, at any stage, confirmed with a tissue biopsy or colorectal polyp/adenoma/mass that is equal or larger than 1 cm in pre-enrollment colonoscopy with residual lesion in the colon of sufficient size to require additional surgical excision or complex colonoscopic polypectomy.
* Subject understands the study procedures and is able to provided informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subject has actively bleeding hemorrhoids (blood on toilet paper or bright red blood clots in the toilet bowel during bowel movement).
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women, 40-90 years of age, inclusive, each with a colonoscopic biopsy-based diagnosis of CRC and/or a pre-malignant colorectal lesion with large enough residual lesion to require subsequent surgical excision or complex colonoscopic polypectomy.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To provide stool and blood specimens to assess new markers for the detection of CRC | 33 months

SECONDARY OUTCOMES:
To provide stool and blood specimens for use as controls when assessing new markers for the detection of neoplasms in other locations within the digestive tract (esophagus, stomach, pancreas, etc.) | 33 months
To provide stool and blood specimens for a biorepository for future cancer-related diagnostic test development | 33 months
To provide quality control material for use in assessing performance of developed assays | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Domanico, Study Chair — Exact Sciences
Locations (22):
- United States (21):
  - John D. Homan, MD, Newport Beach, California
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Gulf Coast Research Group, LLC, Holiday, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Colon and Rectal Surgery Associates, Metairie, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - DBA Boone Hospital Center, Columbia, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Main Line Gastroenterology Associates, Malvern, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Gastro One, Germantown, Tennessee
  - Blue Ridge Medical Researcj, Lynchburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
- Forzani & MacPhali Colon Cancer Screening Centre, Calgary, Alberta, Canada